CLINICAL TRIAL: NCT02985593
Title: A Phase 1, Single-Blind, Randomized, Placebo-Controlled, Single-Dose or Open-Label Multiple-Dose Study of KHK4083 in Healthy Adults and Subjects With Ulcerative Colitis
Brief Title: A Phase 1 Study of KHK4083 in Healthy Volunteers and Subjects With Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4083-003
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Healthy Men and Subjects With Ulcerative Colitis
MeSH Terms: interventions — KHK4083

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KHK4083 (Experimental): IV/SC administration
  Interventions: Drug: KHK4083
- Placebo (Placebo Comparator): IV/SC administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK4083
  Arms: KHK4083
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the safety and tolerability of a single intravenous (IV) or subcutaneous (SC) dose of KHK4083 in Japanese or White healthy men in a placebo-controlled, single-blind comparative study, and to evaluate the safety and tolerability of multiple IV doses of KHK4083 in subjects with ulcerative colitis in an open-label study.

ELIGIBILITY:
"Part1:

Inclusion Criteria:

1. Voluntary written informed consent to participate in the study;
2. Japanese or White men ≥20 and <45 years at the time of informed consent;

Exclusion Criteria:

1. Current illness requiring treatment;
2. Current respiratory, gastric, renal, or liver disease;

Part2:

Inclusion Criteria:

1. Voluntary written informed consent to participate in the study;
2. Men or women ≥20 years of age at the time of informed consent;
3. Ulcerative colitis diagnosed ≥6 months prior to informed consent;
4. Moderate or more severe ulcerative colitis;

Exclusion Criteria:

1. Definitive diagnosis of bacillary dysentery, amebic colitis, Salmonella enteritis, Campylobacter enteritis, colonic tuberculosis, Chlamydia enteritis, Crohn's disease, radiation colitis, drug-induced colitis, angiolymphoid hyperplasia, ischemic colitis, or intestinal Behcet's disease;
2. Any of the following clinically significant concurrent illnesses:

   * Type 1 diabetes
   * Poorly controlled type 2 diabetes (HbA1c >8.5%)
   * Congestive heart failure (class II to IV of the New York Heart Association classification)
   * Myocardial infarction within 1 year
   * Unstable angina pectoris within 1 year
   * Poorly controlled hypertension (systolic pressure >150 mmHg or diastolic pressure >90 mmHg at screening)
   * Severe chronic lung diseases requiring oxygen therapy
   * Multiple sclerosis or other demyelinating diseases
   * Active malignancies, or onset or a history of treatment of malignancies within 5 years prior to informed consent (except for resected or surgically cured epithelial carcinoma of the uterine cervix, cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or ductal carcinoma);
3. Current or past history of clinically significant cardiovascular, liver, renal, respiratory, hematologic, central nervous system, psychiatric, or autoimmune diseases/disorders other than those in 2);
4. Suspected or confirmed symptomatic stenosis of the colon, abdominal abscess, or ischemic colitis based on clinical or radiographic data within 1 year prior to enrollment; suspected or confirmed toxic megacolon or history of toxic megacolon; history of any colonic resection, subtotal or total colectomy, ileostomy, or colostomy; or any previous surgery for ulcerative colitis or an anticipated requirement for surgery for ulcerative colitis;
5. Known colonic dysplasia, adenomas, or polyposis (excluding benign polyposis);
6. Any planned surgical treatment during the study;
7. Clostridium difficile infection within 8 weeks prior to enrollment;
8. Any active infection, including Grade ≥2 localized diseases per Common Terminology Criteria for Adverse Events, version 4.0, Japan Clinical Oncology Group edition (CTCAE v4.0-JCOG), within 4 weeks prior to enrollment;
9. Treatment with 5-aminosalicylic acid (5-ASA) enema, 5-ASA suppository, steroid enema, or steroid suppository within 2 weeks prior to enrollment;
10. Treatment with adalimumab within 2 weeks prior to enrollment or treatment with infliximab within 8 weeks prior to enrollment;

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2017-12-26 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) or drug-related TEAEs and their nature | Part1: Up to 18 weeks post drug administration, Part2: Up to 22 weeks post drug administration

SECONDARY OUTCOMES:
Serum KHK4083 concentration | Part1: Up to 18 weeks post drug administration, Part2: Up to 22 weeks post drug administration
Maximum concentration (Cmax) of KHK4083 | Part1: Up to 18 weeks post drug administration, Part2: Up to 22 weeks post drug administration
Time to reach Cmax (tmax) of KHK4083 | Part1: Up to 18 weeks post drug administration, Part2: Up to 22 weeks post drug administration
Area under the curve (AUC) of KHK4083 | Part1: Up to 18 weeks post drug administration, Part2: Up to 22 weeks post drug administration
Anti-KHK4083 antibody production | art1: Up to 18 weeks post drug administration, Part2: Up to 22 weeks post drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided